CLINICAL TRIAL: NCT06750159
Title: Clinical Study of AKR1B10 for Monitoring Postoperative Recurrence of Hepatocellular Carcinoma
Brief Title: The Use of AKR1B10 for Monitoring Postoperative Recurrence of Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Shunda Du, Head of Liver Surgery Department, Peking Union Medical College Hospital
Other Study IDs: I-24PJ2284
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Residual serum of patients' routine blood tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — no intervention(observational study)

SUMMARY:
Based on the clue that the serum marker AKR1B10 found in the investigators' previous study can be used as an effective indicator for detecting HCC and preHCC, the role and value of AKR1B10 as a new tumor marker for evaluating the recurrence monitoring of HCC after radical surgical resection needs further study, as to provide detailed clinical research data and scientific basis for improving the survival rate of HCC patients.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) is the fourth most common malignancy worldwide and has the second highest mortality rate of all malignancies. Primary liver cancer mainly includes Hepatocellular carcinoma (HCC) and Intrahepatic cholangiocarcinoma (Intrahepatic cholangiocarcinoma). ICC and Combined hepatocellular cholangiocarcinoma (cHCC-CCA) were three different pathologic types. HCC accounts for more than 80% of primary liver cancer cases globally.

Radical hepatocellular carcinoma resection is the main treatment for early HCC, and surgical treatment is the exact way to improve the survival rate. However, the high postoperative recurrence rate seriously affects the prognosis of patients, and the earlier the recurrence, the worse the prognosis. Within 2 years after surgery, it is considered to be the time of early recurrence of hepatocellular carcinoma after surgery, and effective monitoring can remind us of the recurrence of disease in time.

However, at present, there is still a lack of ideal real-time monitoring and diagnostic indicators to evaluate the efficacy of surgical resection and monitor recurrence. At present, postoperative efficacy evaluation and recurrence monitoring of HCC are mainly conducted by means of serological markers (such as alpha-fetoprotein (AFP), abnormal prothrombin (DCP), etc.) combined with imaging examination (such as ultrasound, CT, MRI, etc.) and puncture biopsy. The half-life of AFP in vivo is as long as 6-7 days, so it cannot reflect the residual tumor in vivo in time, and is not suitable for evaluating the efficacy of postoperative resection of HCC and monitoring recurrence. However, the long-term clinical application of DCP has proved that its sensitivity and specificity for liver cancer are not ideal. Therefore, we hope to find a serological marker with higher sensitivity and specificity for HCC, combined with imaging, to accurately evaluate the postoperative efficacy of HCC and monitor recurrence.

AKR1B10 is a monomer reductase that uses homamide adenine dinucleotide phosphate (NADPH) as a coenzyme to catalyze the conversion of endogenous and exogenous carbonyl compounds to alcohol groups, with a half-life of 23 hours in vivo. Under normal circumstances, AKR1B10 is highly expressed in human intestinal tissues, but very low or no expression in liver, lung, breast and other tissues. However, AKR1B10 is highly expressed in hepatocellular carcinoma tissues, and Prof. Cao Deliang cloned AKR1B10 from human primary liver cancer tissues for the first time in 1995. Multiple previous studies have shown that AKR1B10 can be used as a novel marker of primary liver cancer, and its sensitivity and specificity in detecting early liver cancer are significantly better than AFP, in particular, it can sensitively and rapidly reflect the tumor load in vivo, and has functions of liver cancer screening and early diagnosis, which has pioneering significance and great clinical value in the field of liver cancer prevention and treatment. Because AKR1B10 has the characteristics of short half-life and rapid disease changes, postoperative serum AKR1B10 protein detection in patients with liver cancer may be able to know whether tumor cells remain in the body after surgery earlier, providing a scientific basis for doctors to make reasonable postoperative treatment plans, and monitoring possible recurrence during follow-up. However, whether AKR1B10 can be used for efficacy evaluation and recurrence monitoring after radical resection of hepatocellular carcinoma has not been studied and reported.

Based on this, the investigators hypothesized that serum AKR1B10 can provide timely postoperative evaluation and recurrence monitoring after radical resection of hepatocellular carcinoma.

Based on previous studies and real world studies, this study intends to adopt a multicenter, prospective and cohort study, with AKR1B10 expression level as the main observation indicator, combined with existing clinical indicators DCP and AFP, to study the changes of serum AKR1B10, AFP and DCP levels, and evaluate the effect of surgical treatment in HCC patients. At the same time, monitoring the recurrence of HCC is expected to provide a new and reliable method for the evaluation of efficacy and recurrence monitoring after radical resection of HCC, and provide accurate guidance for scientific treatment of HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria of primary hepatocellular carcinoma.
* Meet the criteria for radical resection of hepatocellular carcinoma.
* No anti-cancer treatment before the first diagnosis.

Exclusion Criteria:

* Patients who are pregnant or nursing.
* Patients with incomplete clinical data, serological and imaging findings.
* Patients who were lost to follow-up before the observation endpoint.
* Complicated with serious heart, brain, lung, kidney, hematopoietic and other system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have diagnosed with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
post-operation recurrence or death | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial